CLINICAL TRIAL: NCT01503632
Title: A Comprehensive Approach to Improve Medication Adherence in Pediatric ALL
Brief Title: Assessing Compliance With Mercaptopurine Treatment in Younger Patients With Acute Lymphoblastic Leukemia in First Remission
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ACCL1033; NCI-2012-00105 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S12-01789; CDR0000721559; ACCL1033 (Other: Children's Oncology Group); COG-ACCL1033 (Other: DCP); ACCL1033 (Other: CTEP); R01CA174683 (NIH); U10CA095861 (NIH); UG1CA189955 (NIH); NCT01476852 (obsolete NCT alias)
Record Dates: First submitted 2012-01-03; First posted 2012-01-04 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Behavior Therapy; Mercaptopurine; azathiopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (intervention program and mercaptopurine) (Experimental): See detailed description.
  Interventions: Behavioral: Behavioral Intervention; Behavioral: Compliance Monitoring; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Other: Questionnaire Administration
- Arm II (standard of care and mercaptopurine) (Active Comparator): Patients receive the usual standard of care and the mercaptopurine from the MEMS® medication bottle with TrackCap™ as patients in arm I. Patients and caregivers also view an interactive multimedia educational program on day 29.
  Interventions: Behavioral: Compliance Monitoring; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Other: Questionnaire Administration; Procedure: Standard Follow-Up Care

INTERVENTIONS:
Behavioral: Behavioral Intervention — Receive intervention program
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (intervention program and mercaptopurine)
Behavioral: Compliance Monitoring — Correlative studies
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mercaptopurine — Given orally
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Other: Questionnaire Administration — Ancillary studies
Procedure: Standard Follow-Up Care — Receive usual standard of care
  Arms: Arm II (standard of care and mercaptopurine)

SUMMARY:
This randomized phase III trial studies compliance to a mercaptopurine treatment intervention compared to standard of care in younger patients with acute lymphoblastic leukemia that has had a decrease in or disappearance of signs and symptoms of cancer (remission). Assessing ways to help patients who have acute lymphoblastic leukemia to take their medications as prescribed may help them in taking their medications more consistently and may improve treatment outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the impact of interventions proposed in intervention program (IP) versus (vs.) education alone (EDU) on adherence to oral 6MP (mercaptopurine) in children with acute lymphoblastic leukemia (ALL). Adherence will be measured by: i) Medication Event Monitoring Systems (MEMS) (primary measure of adherence to oral 6MP, providing real-time data; ii) red cell thioguanine nucleotide (TGN) levels (providing data on chronic, systemic 6MP exposure).

SECONDARY OBJECTIVES:

I. Examine the modifying effect of sociodemographic and psychosocial variables, and the mediating effect of health beliefs/ knowledge on change in adherence with intervention.

II. Determine impact of IP vs. EDU on risk of relapse of ALL.

OUTLINE: Patients are randomized to 1 of 2 intervention arms.

ARM I: Patients receive the Patients Supply Kit containing an electronic pill monitoring system, a MEMS® medication bottle with TrackCap™ with standard resistant cap, and written instructions for the patient and pharmacist. Parents and/or caregivers are also trained to supervise patients' intake of the medication. Beginning on day 1, patients start using the MEMS® medication bottle with TrackCap™. Clinical research assistants contact patients and parents by telephone the next day to confirm that TrackCap™ is being used, to identify any obstacles, and to determine solutions. Beginning on day 29, patients and caregivers view an interactive multimedia educational program on-line or via DVD. Patients also receive a customized electronic mercaptopurine schedule and automated customized text message reminders delivered via cellular phone or web-based interface. Patients and caregivers are instructed to return the MEMS® medication bottle with TrackCap™ to the clinic by day 141.

ARM II: Patients receive the usual standard of care and the mercaptopurine from the MEMS® medication bottle with TrackCap™ as patients in arm I. Patients and caregivers also view an interactive multimedia educational program on day 29.

After completion of study treatment, patients are followed up every 6 months for 5 years and then annually until 10 years from diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALL, in first remission; enrollment on a Children Oncology Group (COG) therapeutic study for ALL is not required
* At the time of enrollment, patient must have completed at least 24 weeks of maintenance chemotherapy, and is scheduled to receive at least 24 more weeks of maintenance chemotherapy
* Receiving continuous oral 6MP during the maintenance phase of therapy for ALL (held only for toxicity or illness), and will be returning to the clinic every 4 weeks for scheduled appointments while enrolled on COG ACCL1033 (between days 1 and 141)
* Has a designated parent or caregiver who is willing to enter into a mutual agreement with the patient to participate in a daily supervised medication administration routine
* Able and willing to use the MEMS® TrackCap™ (e.g., not using a pillbox or prescribed liquid 6MP)
* Parent/caregiver and patient (if 12 years and older) must be willing to use a cellular telephone to receive medication reminders via text messaging during study period
* Patient and parent/caregiver must speak English or Spanish
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with Down syndrome
* Patients who previously participated in or are currently participating in another intervention clinical trial designed to improve adherence

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 570 (Actual)
Dates: Start 2012-02-21 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with adherence rate greater than or equal to 95% to mercaptopurine as measured by MEMS® | 4 months
  Compared between the IP and EDU groups using logistic regression. Mercaptopurine levels will be modeled as a function of time to examine longitudinal changes to 6TGN levels between the treatment groups using the generalized estimating equation (GEE) method for longitudinal normally distributed data.
Proportion of patients with adherence rate greater than or equal to 95% to mercaptopurine as measured by red cell TGN levels | 4 months
  Compared between the IP and EDU groups using logistic regression. Mercaptopurine levels will be modeled as a function of time to examine longitudinal changes to 6TGN levels between the treatment groups using the GEE method for longitudinal normally distributed data.

SECONDARY OUTCOMES:
Proportion of adherence patients by sociodemographic and psychosocial variables | 4 months
  Evaluated analytically by logistic regression methods.
Mediating effect of health beliefs/ knowledge on change in adherence with intervention | 4 months
  Evaluated analytically by logistic regression methods.
Impact of IP vs. EDU on risk of relapse in children with ALL | Up to 10 years
  An intention-to-treat analysis will be used to compare the effectiveness of EDU and IP interventions in decreasing the risk of relapse. Cox proportional hazards regression models will be used to examine the impact of intervention on relapse. Covariates in the analysis will include clinical and sociodemographic predictors, and the intervention arm (IP vs. EDU).

CONTACTS AND LOCATIONS:
Overall Officials: Smita Bhatia, Principal Investigator — Children's Oncology Group
Locations (102):
- United States (100):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Vannie Cook Children's Clinic, McAllen, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] Bhatia S, Hageman L, Chen Y, Wong FL, McQuaid EL, Duncan C, Mascarenhas L, Freyer D, Mba N, Aristizabal P, Walterhouse D, Lew G, Kempert PH, Russell TB, McNall-Knapp RY, Jacobs S, Dang H, Raetz E, Relling MV, Landier W. Effect of a Daily Text Messaging and Directly Supervised Therapy Intervention on Oral Mercaptopurine Adherence in Children With Acute Lymphoblastic Leukemia: A Randomized Clinical Trial. JAMA Netw Open. 2020 Aug 3;3(8):e2014205. doi: 10.1001/jamanetworkopen.2020.14205. PMID 32852553